CLINICAL TRIAL: NCT06872281
Title: A Randomized Controlled Trial Comparing Fractional Bipolar Radiofrequency Therapy VS Sham for Treatment of Vaginal Laxity in Premenopausal Women
Brief Title: Fractional Bipolar Radiofrequency Therapy VS Sham for Treatment of Vaginal Laxity in Premenopausal Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: InMode MD Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COA.No. MURA2025/130
Record Dates: First submitted 2025-02-17; First posted 2025-03-12 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Vaginal Laxity
Keywords: fractional bipolar radiofrequency therapy

STUDY DESIGN:
Intervention Model Description: Treatment was performed using the Empower RF Morpheus8V device (InMode),
  * Insert device into vaginal
  * Do not need for anesthesia
  * Applying fractional bipolar RF energy in a stamping method
  * 50% overlap along the entire length of the vagina to the introitus, At intervals of 9, 10:30, 12, 1:30, 3, 4:30, 6, and 7:30.
  * Two passes were made at depths of 1, 2, and 3 mm.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: This study employs a double-blind design to minimize bias by blinding both the patients and evaluators. All patients, regardless of group, will remain blinded. The sham group will receive treatment with a specialized sham device that mimics the treatment group's equipment. There are no differences in the design of the tip device, the auditory signal (beeping), or the pulse count display. The physician managing the allocation, will not be involved in the treatment procedures or the assessment process. Subjective outcomes, such as questionnaires (VLQ, FSFI, FGSIS, ICIG-VS, PGI-I), will be assessed by a research assistant from the urogynecology clinic who is blinded to the group assignments, ensuring she is unaware of which patients received the actual treatment and which received the sham.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intervention (fractional bipolar radiofrequency therapy) (Active Comparator): A single treatment with intravaginal device for fractional bipolar radiofrequency therapy. Using the EmpowerRF platform with the Morpheus8V applicator, RF energy was applied via 24 microneedles, to release the radiofrequency energy to the vaginal mucosa
  Interventions: Device: Fractional bipolar radiofrequency
- Sham group (Sham Comparator): The sham group will receive treatment with a specialized sham device that mimics the treatment group's equipment. There are no differences in the design of the tip device, the auditory signal (beeping), or the pulse count display.
  Interventions: Device: Sham device

INTERVENTIONS:
Device: Fractional bipolar radiofrequency — The treatment group will receive a single treatment of intravaginal fractional bipolar radiofrequency therapy.
  Arms: Intervention (fractional bipolar radiofrequency therapy)
Device: Sham device — The sham group will receive treatment with a specialized sham device that mimics the treatment group's equipment. There are no differences in the design of the tip device, the auditory signal (beeping), or the pulse count display.
  Arms: Sham group

SUMMARY:
Knowledge gap: Lack of randomized controlled trials evaluating the efficacy of fractional bipolar radiofrequency therapy compared to a sham treatment for vaginal laxity in premenopausal women.

Primary outcomes

* Subjective outcomes: The Vaginal Laxity Questionnaire (VLQ) Secondary outcomes
* Subjective outcomes

  * The Thai version of the Female Sexual Function Index (FSFI) will be administered to evaluate sexual function.
  * The Thai version of the Female Genital Self-Image Scale (FGSIS)
  * The International Consultation on Incontinence Questionnaire-Vaginal Symptoms (ICIQ-VS), validated in Thai
  * The Patient Global Impression of Improvement (PGI-I)
  * Patients will report any side effects or adverse events experienced during the study.
* Objective outcomes - Vaginal wall thickness will be assessed using 3D transvaginal ultrasound imaging, following the standardized protocol established in previous studies.

PICO:

P (Population): Premenopausal women with clinically diagnosed vaginal laxity who are sexually active.

I (Intervention): Fractional bipolar radiofrequency therapy (single treatment)

C (Comparison): Sham treatment (placebo).

O (Outcomes):

* Primary Outcome: Improvement in vaginal laxity as assessed by the Vaginal Laxity Questionnaire (VLQ).
* Secondary Outcomes: Patient satisfaction with treatment (measured by the Patient Global Impression of Improvement - PGI-I)., Changes in sexual function (assessed using the Thai version of the Female Sexual Function Index - FSFI).

Perception of genital self-image (evaluated using the Thai version of the Female Genital Self-Image Scale - FGSIS)., Evaluation of vaginal symptoms (using the International Consultation on Incontinence Questionnaire-Vaginal Symptoms - ICIQ-VS), Objective assessment of vaginal wall thickness through 3D transvaginal ultrasound, Recording of any side effects or adverse events associated with the treatment.

Study Design:

A double-blind, randomized controlled trial (RCT) conducted at the Female Pelvic Medicine and Reconstructive Surgery clinic in Ramathibodi Hospital.

DETAILED DESCRIPTION:
Vaginal laxity is a prevalent concern among premenopausal women today. A retrospective cohort study found that 24% of women reported experiencing vaginal laxity. According to the IUGA/ICS 2018 definition, vaginal laxity is characterized by a sensation of looseness in the vagina.

Fractional bipolar radiofrequency therapy has emerged as a promising minimally invasive treatment modality. This non-ablative approach uses fractional RF technology with microneedles to deliver thermal injury to the subdermis, stimulating collagen production, promoting tissue remodeling and improving tissue tightening, potentially addressing symptoms associated with vaginal laxity. Recent advancements in RF technology have led to its increasing use in aesthetic and gynecological applications. Evidence suggests that RF microneedling effectively remodels subdermal fat and improves skin firmness. However, no previous study has been conducted on the treatment of vaginal laxity using fractional bipolar radiofrequency (with microneedling), highlighting the need for rigorous scientific evaluation to provide conclusive evidence on its effectiveness, including improvements in sexual function and safety.

Additionally, the use of 3D transvaginal ultrasound to measure vaginal wall thickness is still limited in clinical studies. It is necessary to investigate whether fractional bipolar radiofrequency can improve vaginal wall thickness and explore the association between vaginal wall thickness and the clinical presentation of vaginal laxity in patients.

This study aims to address this gap by conducting a first randomized controlled trial to compare the efficacy of fractional bipolar radiofrequency therapy with a sham treatment in premenopausal women. By employing a methodological approach, this research seeks to contribute valuable insights into the clinical benefits of fractional bipolar radiofrequency therapy, ultimately guiding future treatment strategies for vaginal laxity.

Primary Objective:

- To evaluate and compare the efficacy of fractional bipolar radiofrequency therapy versus a sham treatment for vaginal laxity in premenopausal women.

Secondary Objectives (if any):

* To evaluate patient satisfaction and changes in sexual function before and after fractional bipolar radiofrequency therapy VS sham treatment.
* To assess alterations in vaginal thickness based on 3D transvaginal ultrasound before and after fractional bipolar radiofrequency therapy Vs sham treatment.
* To evaluate any potential side effects or adverse events associated with intravaginal fractional bipolar radiofrequency therapy.

Study design/methodology:

* Study design: A double-blind, randomized controlled trial
* Study Population: Premenopausal women with clinically diagnosed vaginal laxity who are sexually active.

Specifications of Fractional Radiofrequency energy (Morpheus8V from Inmode company)

* Configuration: 24 gold coated micropins
* Depth profile: 1-3 mm
* Pin profile: 300um diameter with insulated 0.5 mm conductive tip
* Treatment depth: operator adjustable
* Principle: Microneedling with fractional RF: delivery RF energy to depths from 0.5-3.5 mm below the surface, induced additional thermal stimulation, superior neo-collagenesis than with RF energy alone
* Treatment was performed using the Empower RF Morpheus8V device (InMode), applying fractional bipolar RF energy in a stamping method with 50% overlap along the entire length of the vagina to the introitus, at intervals of 9, 10:30, 12, 1:30, 3, 4:30, 6, and 7:30.
* Two passes were made at depths of 1, 2, and 3 mm.

Participant timeline and Procedures:

Week 0:

* Screening and enrollment, Eligibility screening, Inform consent, General advice for PFMT
* Baseline assessment: Demographic data, Questionnaires (VLQ, FSFI, FGSIS, ICIQ-VS)
* Physical examination: PV: Evaluate genital hiatus (Gh), vaginal caliber
* 3D endovaginal US: Evaluate baseline vaginal thickness.

Week 1

* Intervention *Radiofrequency therapy VS Sham 72 hours post-intervention:
* Telemedicine Inquire with the patients about any adverse events they may have experienced following the intervention

Week 4 (1-month post-intervention):

- Telemedicine/questionnaires by mail Questionnaires (VLQ, FSFI, FGSIS, ICIQ-VS), Assessment for any adverse events, The Patient Global Impression of Improvement (PGI-I)

Week 13 (3 months post-intervention):

* Follow-up visit Questionnaires (VLQ, FSFI, FGSIS, ICIQ-VS)
* Assessment for any adverse events
* The Patient Global Impression of Improvement (PGI-I)
* Physical examination PV: Evaluate genital hiatus (Gh), vaginal caliber
* 3D endovaginal US Evaluate vaginal thickness post-RF treatment

Discontinuation/withdrawal criteria:

* Adverse Events: Development of serious adverse effects or complications related to the therapy, such as severe pain, infection, or significant bleeding. Or any signs or concerns that the participant might not be safe to continue, as determined by the investigator.
* Pregnancy: If a participant becomes pregnant during the study, they may need to withdraw to ensure safety for both the mother and the fetus.
* Medical Conditions: Emergence of new medical conditions or exacerbation of existing conditions that could complicate participation or the study's objectives such as active genital infection.
* Patient Preference: Participant's decision to withdraw from the study for personal reasons, including dissatisfaction with the treatment or its effects.

Adverse Event Reporting:

* Pain, discomfort, or a burning sensation during or after the procedure.
* Worsening of urinary symptoms
* The presence of vaginal burn
* Vaginal discharge
* The presence of abnormal vaginal bleeding (spotting).
* Swelling and bruising: Mild to moderate swelling and bruising at the treatment site
* Infection: There is a small risk of infection at the site of microneedling if proper post-treatment care is not followed.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women
* Age 20-55 years
* Reported symptoms of vaginal looseness with a score of at least 1 on The Vaginal Laxity Questionnaire (VLQ)
* Sexually active (≥1 time/month)
* Willing to undergo vaginal energy-based treatment and attend follow-up visits 3 months after treatment

Exclusion Criteria:

* - Presence of sexually transmitted diseases or active genital lesions
* Currently pregnant or planning for conception during study period
* Pelvic organ prolapse (POP ≥ Stage II)
* Previous treatment for vaginal laxity with modalities other than pelvic floor muscle training
* Currently using intrauterine devices for contraception
* Presence of any active electrical implant such as pacemaker, internal defibrillator
* Current condition of genital cancer

Ages: 20 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 56 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
The Vaginal Laxity Questionnaire (VLQ) | From enrollment to the end of treatment at 12 weeks
  Subjective outcomes
  * The Vaginal Laxity Questionnaire (VLQ) will be used to assess patient-reported vaginal laxity.
  * A score of 1-3 indicates positive for vaginal laxity (1 = severe, 2 = moderate, 3 = mild symptom).
  * A score of 4-7 indicates no vaginal laxity, with 7 representing the greatest vaginal tightness.
  * A higher VLQ score post-treatment reflects improvement in vaginal laxity.

SECONDARY OUTCOMES:
Subjective outcomes: The Patient Global Impression of Improvement (PGI-I) | From 4-week post-treatment to the end of the 12-week treatment period
  The Patient Global Impression of Improvement (PGI-I) will measure overall patient satisfaction with treatment outcomes. It is a global index used to assess the response of vaginal laxity to therapy. The PGI-I is a single-question transition scale asking patients to rate their vaginal laxity condition compared to before treatment, on a scale from 1 (very much better) to 7 (very much worse).
Subjective outcome: Patient-reported adverse events | From post-treatment to the end of the 12-week treatment period
  Patients will report any side effects or adverse events experienced during the study.
  * Pain or discomfort will be assessed using "a visual analog scale" from 0 to 10 (0 = no pain, 10 = worst pain).
  * Other adverse events, such as abnormal vaginal bleeding, abnormal vaginal discharge, vaginal burning sensation, and dyspareunia, will be reported as yes (if present) or no (if not present)
Subjective outcome: The Thai version of the Female Sexual Function Index (FSFI) | From enrollment to the end of treatment at 12 weeks
  The FSFI comprises of a 19-item questionnaire focused on sexual functioning. There are 6 domain scores (desire, arousal, lubrication, orgasm, satisfaction, pain) belonging to the FSFI and that are summed to obtain the overall score.
  The rule of thumb for the overall result is that scores equal to or below 26.55 are classed as indicating female sexual dysfunction (FSD).
  The domain scores are derived from the multiplication of the sum of domain items points and the domain factor. By adding the six domains, the final result can be obtained.
  Usually, for domains in which the score is zero, this is indicative of the subject having reported there was no sexual activity during the past 4 weeks.
Subjective outcome: The Thai version of the Female Genital Self-Image Scale (FGSIS) | From enrollment to the end of treatment at 12 weeks
  The FGSIS score stands for the Female Genital Self-Image Scale. It is used to assess how women perceive their genitalia and can provide insight into their satisfaction, body image, and how these factors may impact sexual function and health-related quality of life.
  The FGSIS includes a series of statements or questions, usually answered on a 4-point or 5-point Likert scale, with responses such as:
  * Strongly Disagree
  * Disagree
  * Neutral
  * Agree
  * Strongly Agree
  Total Score:
  • The responses are totaled to give an overall score.
  Interpretation of Scores:
  * Low Scores: These suggest a more negative or dissatisfied genital self-image. This may reflect concerns or dissatisfaction with the appearance, function, or health of the genital area, which could be related to emotional or sexual concerns.
  * High Scores: Higher scores indicate a more positive or satisfied genital self-image, suggesting greater confidence or comfort with one's body in this regard.
Subjective outcome: The International Consultation on Incontinence Questionnaire-Vaginal Symptoms (ICIQ-VS) | From enrollment to the end of treatment at 12 weeks
  It is a Thai-validated tool used to assess vaginal symptoms, their impact on quality of life, and sexual matters in women.
  Scoring: Each item in the ICIQ-VS is scored on a Likert scale based on severity (e.g., not at all, slightly, moderately, a lot) or frequency (never, sometimes, always). The questionnaire generates a total score as well as scores for each section (vaginal symptoms subscore, quality of life Impact subscore, sexual matters subscore)
  Interpretation of Scores:
  * Low Scores: Suggest minimal or no symptoms, indicating little to no impact on vaginal health, quality of life, or sexual function.
  * High Scores: Suggest more severe symptoms, with greater impact on vaginal health, daily activities, emotional well-being, and sexual satisfaction. A high score indicates that vaginal symptoms are significantly affecting quality of life and sexual function.
Objective outcomes: the difference of vaginal wall thickness before and after intervention | From enrollment to the end of treatment at 12 weeks
  - Vaginal wall thickness will be assessed using 3D transvaginal ultrasound imaging, following the standardized protocol established in previous studies.

CONTACTS AND LOCATIONS:
Overall Officials: Suthanud Premchit, MD, Principal Investigator — Ramathibodi Hospital
Locations (1):
- Faculty of Medicine Ramathibodi Hospital, Mahidol University, Ratchathewi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
Information will be shared in de-identified data.
  Research collaborators will have access to the data.
  Specify that data shared with collaborators will be used for conducting analyses relevant to the study objectives, secondary analyses, or other agreed-upon purposes.
  Data will be shared via a secure institutional repository accessible to collaborators through data-sharing agreements.

REFERENCES:
- [Result] Abdelaziz A, Blusewicz TA, Coley KP, Karram M. Safety, tolerability and short-term efficacy of transvaginal fractional bipolar radiofrequency therapy for symptoms of stress and or mixed incontinence in conjunction with genitourinary syndrome of menopause. Neurourol Urodyn. 2023 Apr;42(4):807-813. doi: 10.1002/nau.25170. Epub 2023 Mar 4. PMID 36870045
- [Result] Millheiser LS, Pauls RN, Herbst SJ, Chen BH. Radiofrequency treatment of vaginal laxity after vaginal delivery: nonsurgical vaginal tightening. J Sex Med. 2010 Sep;7(9):3088-95. doi: 10.1111/j.1743-6109.2010.01910.x. PMID 20584127
- [Result] Wattanakrai P, Limpjaroenviriyakul N, Thongtan D, Wattanayingcharoenchai R, Manonai J. The efficacy and safety of a combined multipolar radiofrequency with pulsed electromagnetic field technology for the treatment of vaginal laxity: a double-blinded, randomized, sham-controlled trial. Lasers Med Sci. 2022 Apr;37(3):1829-1842. doi: 10.1007/s10103-021-03438-3. Epub 2021 Oct 14. PMID 34647191
- [Result] Polland A, Duong V, Furuya R, Fitzgerald JJ, Wang H, Iwamoto A, Bradley S, Iglesia CB. Description of Vaginal Laxity and Prolapse and Correlation With Sexual Function (DeVeLoPS). Sex Med. 2021 Dec;9(6):100443. doi: 10.1016/j.esxm.2021.100443. Epub 2021 Oct 8. PMID 34629323
- [Result] Dayan E. Noninvasive Vulvar and Intravaginal Treatments. Clin Plast Surg. 2022 Oct;49(4):505-508. doi: 10.1016/j.cps.2022.07.004. PMID 36162945
- [Result] Krychman ML. Vaginal Laxity Issues, Answers and Implications for Female Sexual Function. J Sex Med. 2016 Oct;13(10):1445-7. doi: 10.1016/j.jsxm.2016.07.016. Epub 2016 Aug 23. No abstract available. PMID 27567072

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-14): https://cdn.clinicaltrials.gov/large-docs/81/NCT06872281/Prot_SAP_000.pdf